CLINICAL TRIAL: NCT07406230
Title: Methotrexate Early Toxicity Monitoring in Primary Central Nervous System Lymphomas (PCNSL)
Brief Title: Methotrexate Early Toxicity Monitoring
Acronym: METoxiM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM24_0313; ID RCB: 2025-A01802-47 (Other: ANSM)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Primary Central Nervous System Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients suffering from primary central nervous system lymphomas PCNSL (Experimental)
  Interventions: Other: methotrexate plasmatic dosing

INTERVENTIONS:
Other: methotrexate plasmatic dosing — Methotrexate (MTX) dosage at 2,4,6,8,24 and 48 hours

SUMMARY:
High-dose methotrexate (MTX) is the main componement of first line treatment in primary central nervous system lymphoma. Renal toxicity is the main dose limiting toxicity because of major MTX elimination by the kidneys. MTX crystallizes in renal tubules, leading to a renal failure (RF) and further delaying its elimination. When RF occurs, MTX accumulates, prolonging the duration of treatment exposure. MTX prolonging exposure can cause life-threatening complications and delay further treatments in the patient. Preventive measures have been developped, such as alkaline fluid hyperhydration and folic acid administration, to try to reduce the risk of these adverse events.

In suspected severe RF in link to MTX is suspected, glucarpidase can be administared. However, this is an expensive treatment and not all patients recover normal renal function despite its use.

MTX is an essential treatment for the management of PCNSL which is currently a curable disease especially in patients who are able to receive a consolidation treatment as thiotepa-based intensive consolidation followed by autologous stem cell transplantation (IC-ASCT). IC-ASCT requires a normal renal function, which could be impaired by severe RF secondary to MTX.

The purpose of the study is to investigate how early dosing MTX could be used to simulate late concentrations. Early monitoring of MTX elimination could be implemented to identify patients at risk of delayed elimination and thus introduce rapid mesures as early administration of glucarpidase.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 years or older,
* Patient with a primary lymphoma of the central nervous system, histologically or cytologically proven,
* Patient eligible for high-dose methotrexate treatment (> at 500 mg/m 2), in the first line of treatment,
* Patient who has received information regarding the study and signed an informed consent,
* Patient beneficiary or entitled to a social security scheme.

Exclusion Criteria:

* Patient treated with a therapy complementary to the standard 1st-line treatment based on high-dose MTX as part of a clinical research protocol,
* Patient in a period of exclusion from another research protocol at the time of signing consent,
* Subjects covered by articles L1121-5 to 1121-8 of the Public Health Code (minor patient, adult patient under guardianship or curatorship, patient deprived of liberty, pregnant or breastfeeding woman).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy measurement of Bayesian model | 48 hours post MTX
  Determine, in patients with Primary Central Nervous System Lymphoma (PCNL), the most efficient Bayesian model for predicting the delay in MTX elimination using a pharmacometry approach (in silico modeling based on a population approach) based on the early dosage of methotrexate in plasma.

SECONDARY OUTCOMES:
Determine the Bayesian model for predicting renal toxicity of MTX T48H using a pharmacometric approach (in silico modeling) based on early dosing of methotrexate in plasma | 48 hours post MTX
  Renal toxicity shall be defined as acute renal failure graded according to CTCAE V5 in relation to the value of serum creatinine before administration of MTX.
Determine the bayesian model for predicting MTX clearance 72 hours after MTX using a pharmacometric approach (in silico modeling) based on early dosing of methotrexate in plasma | 72 hours post MTX
  Delay in elimination will be defined by a methotrexate dosage 72 hours after administration (T72H) beyond 0.2 μmol/L.
Estimate in an exploratory approach the performance of the Bayesian model for predicting the delay in MTX elimination at 48 hours using a pharmacometric approach (in silico modeling) | 48 hours post
  Correlation between, early dosage of methotrexate in plasma and other parameters of interest measured at baseline (before MTX administration) such as patient age, albumin and creatinine clearance.
Estimate in an exploratory approach the performance of the Bayesian model for predicting overexposure to MTX at 48 hours using a pharmacometric approach (in silico modeling) | 48 hours post MTX
  Correlation between, early dosage of methotrexate in plasma and other parameters of interest measured at baseline (before MTX administration) such as patient age, albumin and creatinine clearance. Overexposure to MTX is defined by a measured T48H > 10 μmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: François Crémieux, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France